CLINICAL TRIAL: NCT04438070
Title: COVID Screening Strategies in Homeless Shelters
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: St. Joseph's Healthcare Hamilton (Other)
Collaborators: Timothy O'Shea (Unknown); Marek Smieja (Unknown); Lawrence Mbuagbaw (Unknown)
Responsible Party: Principal Investigator, Marek Smieja, Principal Investigator, St. Joseph's Healthcare Hamilton
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: 2020-10864-T
Record Dates: First submitted 2020-06-17; First posted 2020-06-18 (Actual); Last update posted 2020-06-18 (Actual); Status verified 2020-06

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Intervention Model Description: Cluster randomized multi-center trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Daily active screening only (Placebo Comparator)
  Interventions: Diagnostic Test: COVID-19 Swab
- Daily active screening and self-collected nasal swab (Experimental)
  Interventions: Diagnostic Test: COVID-19 Swab
- Daily active screening and self-collected oral-nasal swab (Experimental)
  Interventions: Diagnostic Test: COVID-19 Swab
- Daily active screening and nurse collected nasopharyngeal swab (Experimental)
  Interventions: Diagnostic Test: COVID-19 Swab

INTERVENTIONS:
Diagnostic Test: COVID-19 Swab — Nasal, Oral-Nasal combined or Nasopharyngeal swab

SUMMARY:
Residents in homeless shelters will be randomized to 4 different COVID-19 screening strategies with the primary outcome being COVID-19 detection rate.

ELIGIBILITY:
Inclusion Criteria:

* Age greater than or equal to 18
* Able to provide oral consent
* Able to perform a self-collected swab if in the relevant intervention arm

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2020-04-10 (Actual); Primary Completion 2020-06 (Estimated); Study Completion 2020-06 (Estimated)

PRIMARY OUTCOMES:
COVID-19 Detection Rate | 8 weeks

SECONDARY OUTCOMES:
Number of outbreaks | 8 weeks
Enrollment over time | 8 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Various Homeless Shelters, Hamilton, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Mokashi V, Gilchrist J, Smieja N, Maciejewski J, Marttala S, Beal K, Mbuagbaw L, Bulir D, Smieja M, O'Shea T. Four COVID-19 screening strategies for early case identification within the homeless shelter population: a cluster randomized controlled trial. BMC Infect Dis. 2024 Dec 28;24(1):1478. doi: 10.1186/s12879-024-10148-y. PMID 39732649
- [Derived] O'Shea T, Mbuagbaw L, Mokashi V, Bulir D, Gilchrist J, Smieja N, Chong S, Marttala S, Vera V, Cvetkovic A, Smieja M. Comparison of four COVID-19 screening strategies to facilitate early case identification within the homeless shelter population: A structured summary of a study protocol for a randomised controlled trial. Trials. 2020 Nov 23;21(1):941. doi: 10.1186/s13063-020-04890-2. PMID 33225995